CLINICAL TRIAL: NCT01772251
Title: A Single-Center, Multiple-dose, Randomized, Cross-Over, Double-Blind, Placebo-Controlled Study to Evaluate the Pharmacodynamics, Safety, and Tolerability of Oshadi Icp In Patients With Type 1 Diabetes Mellitus - Phase Ib Clinical Study
Brief Title: Safety and Tolerability of Oshadi Icp In Patients With Type 1 Diabetes Mellitus - Phase Ib Clinical Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oshadi Drug Administration (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OS-ICP-P1b-01; 2012-004270-26 (EudraCT Number)
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes Mellitus, Insulin-Dependent, 1
Keywords: Diabetes Mellitus; Oral Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oshadi Icp & placebo (Experimental)
  Interventions: Drug: Oshadi Icp

INTERVENTIONS:
Drug: Oshadi Icp
  Other Names: Oral insulin

SUMMARY:
Diabetes mellitus (DM) is a chronic disease of carbohydrate, fat, and protein metabolism caused by an absolute or relative deficiency of insulin, an anabolic hormone. The current methods of insulin therapy for diabetic patients are multiple daily injection therapy and continuous subcutaneous insulin infusion with an external pump. This rout of administration may lead to hyperinsulinemia as insulin is administered in a non physiological way, targeting mainly extra hepatic tissues (muscle, fat).

A method of providing insulin without the need for injections has been a goal in drug delivery.

Oshadi Drug Administration Ltd. has developed oral carrier for proteins based on biochemistry and quantum theory of biochemical reactions. The carrier enables the absorption of proteins from the gastrointestinal tract in their full structure. Oshadi has also developed the Oshadi Icp - insulin, proinsulin and C-peptide in Oshadi carrier, administrated orally. This study was design in order to evaluate the safety and feasibility of multiple administration of Oshadi Icp

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (according to ADA criteria) for more than 1 year.
* Male/female 18 years old and older.
* BMI≥18.5 and ≤25
* Female of childbearing age must commit to avoid pregnancy and use contraception during the study.
* Patients must understand and be willing to give written informed consent prior to any study procedures or evaluations and be willing to adhere to all study schedules and requirements.

Exclusion Criteria:

* Any history of significant cardiac, renal, neurologic, metabolic, pulmonary, gastrointestinal, hematologic abnormality, chronic hepatic disease or any other disease which in the judgment of the investigator would interfere with the study or confound the results.
* Symptomatic DKA in the last 6 months
* Patients with positive HIV or HCV serology or positive HBsAg at screening.
* History or evidence of any active liver disease.
* History of epilepsy.
* One hypoglycemic seizure episode in the last six months or more than one hypoglycemic seizure episode in the last year.
* History of sever recurrent hypoglycemic unawareness.
* C-peptide >3 mg/ml (fasting)
* Total average daily insulin dosage ≥1 IU/kg of body weight.
* Polycystic ovary syndrome
* Acanthosis nigricans
* 6.5% > HbA1c or HbA1c >10%
* eGFR<60.
* Female patients who are breastfeeding or have a positive pregnancy test at screening or at any time during the study and not willing to practice birth control during study period.
* Inability to give written informed consent
* History of alcohol or drug abuse within 6 months of screening.
* Patients who have a positive urine drug screen for substances of abuse (benzodiazepine, THC, opiates, amphetamines, cocaine) at the screening.
* Mental disorders.
* Patients with poor venous access
* Significant swallowing disorders
* Digestive disorders
* Small bowel surgery
* Any intercurrent disease during the last week prior to screening which in the judgment of the investigator might affect blood glucose level.
* Any infectious disease developed during the 4 weeks prior to the study.
* Malabsorption disorders.
* Any significant abnormality by principal investigator in the baseline laboratory evaluation: liver and kidney functions, electrolytes, albumin, lipase, TSH, hemoglobin, white blood cell count and differential, platelets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events occurence | last follow-up visit (day 23)

SECONDARY OUTCOMES:
• To assess the pharmacodynamic effect of multiple doses of Oshadi Icp as measured by the area under the glucose concentration-time curve | last administration day (day 17)

OTHER OUTCOMES:
• Evaluating the total daily injected insulin dose during administration of Oshadi Icp vs. placebo | Last administration day (day 17)

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel